CLINICAL TRIAL: NCT01552889
Title: Randomized Controlled Trial of Screening for Depression in Cardiac Outpatients
Brief Title: Depression Outpatient Cardiology Screening Study
Acronym: DOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Carney, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201105510
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Depression; Coronary Heart Disease
MeSH Terms: conditions — Depression; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (UC) (No Intervention): Patients will receive only the care provided by their primary care physicians or other medical professionals outside of the study.
- Collaborative Care (CC) (Experimental): Patients randomized to the Collaborate Care (CC) arm of this study will receive brief screening, consultative, and referral services. This collaborative approach includes the patient, the patient's PCP, the cardiologist, and the nurse case manager (NCM), using evidence based recommendations for depression treatment and follow-up care.
  Interventions: Behavioral: Collaborative Care

INTERVENTIONS:
Behavioral: Collaborative Care — No direct treatment will be offered. We will make treatment recommendations to the patient, PCP and cardiologist. Referral to mental health specialist is also possible, depending on need. The nurse case manager will monitor treatment progress and patient status for duration of the intervention period.
  Arms: Collaborative Care (CC)

SUMMARY:
This study compares the effects of depression screening and case management to usual care in cardiology outpatients with documented evidence of coronary heart disease. Despite strong evidence that depression is a risk factor for cardiac events, there is insufficient evidence to support the use of depression screening in cardiac patients.

DETAILED DESCRIPTION:
Depression and cardiovascular disease are highly comorbid, and depression is a risk factor for psychosocial morbidity, poor adherence to medical treatment regimens, physical inactivity, poor physical functioning, and medical morbidity and mortality in cardiac patients, especially following an acute coronary syndrome (ACS). The American Heart Association recently recommended that all cardiac patients be screened for depression in order to improve identification and treatment of this risk factor.

Patients are screened for depression during an outpatient cardiology visit and those that screen positive will be contacted for enrollment into this study. Patients are then randomized to receive collaborative care involving the patient, the patient's primary care physician (PCP), the cardiologist and the nurse case manager, or usual care (the patient is informed he/she screened positive for depression and is advised to contact their PCP and/or cardiologist). The PCP and/or cardiologist are free to evaluate, treat and refer that patient to mental health services as they deem necessary.

Patients in both groups will be monitored for depression severity and duration at 3, 6 and 12 months after enrollment. The course of their depression since enrollment or last follow-up includes remissions, new onsets, relapses, recurrences, and treatment will be determined.

ELIGIBILITY:
Inclusion Criteria:

* recent history of Acute Coronary Syndrome or other cardiac event or documented heart disease
* score of 10 or higher on the Patient Health Questionnaire

Exclusion Criteria:

* suicidal ideation or behavior
* cognitive impairment or inability to read or speak English
* schizophrenia, bipolar disorder
* active substance abuse or alcoholism
* severe valvular disease, severe congestive heart failure, malignancy
* physical limitations that would interfere with participation in the study
* medical contraindications to the use of available antidepressants
* participation in a competing research protocol
* physician or patient refusal

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Carney, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Behavioral Medicine Center at Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care (UC) | Collaborative Care (CC)
Started | 101 | 100
Completed | 90 | 95
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Collaborative Care (CC) | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 64 | 122
  >=65 years | 43 | 36 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.0) | 63.0 (9.5) | 63.05 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 47 | 84
  Male | 64 | 53 | 117
Region of Enrollment [Number; unit: participants]
  United States | 101 | 100 | 201

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory 2
Description: Self report depression symptom inventory. Scale ranges from 0-63. The higher the score the more depression symptoms. A score of 12 or greater is considered to indicate a clinically significant depression.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care (UC) | Collaborative Care (CC)
Number analyzed (Participants) | 101 | 100
units on a scale | 17.4 (9.0) | 15.9 (8.8)

2. Secondary Outcome: Treatment Satisfaction Scale.
Description: This one item scale asks patients to rate their satisfaction with their depression treatment on a one (very dissatisfied) to 5 (very satisfied) scale.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care; Collaborative Care: Same as above
Arm/Group | Usual Care | Collaborative Care
Number analyzed (Participants) | 101 | 100
units on a scale | 3.3 (1.3) | 4.0 (1.1)

3. Secondary Outcome: PROMIS Physical Functioning Scale 10a Short Form
Description: This is a 10 item questionnaire that assesses the respondent's ability to perform common physical activities as rated on a 1-5 scale. The total score is converted to a T score which expresses where the individual ranks relative to the reference group.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Collaborative Care
Number analyzed (Participants) | 101 | 100
units on a scale | 39.6 (4.9) | 39.2 (4.5)

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Usual Care (UC) | Collaborative Care (CC)
All-Cause Mortality (participants affected / at risk) | 8/101 | 1/100
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100
Other Adverse Events (participants affected / at risk) | 0/101 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No